CLINICAL TRIAL: NCT06334497
Title: Letermovir/Valganciclovir Combination Versus Valganciclovir Monotherapy for Treatment of Cytomegalovirus (CMV) Infections in Kidney Transplant Recipients
Brief Title: Letermovir-based Dual Therapy for Treatment of Cytomegalovirus Infections
Acronym: LUCY-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220791; 2023-506216-40-00 (Other: EU CT)
Record Dates: First submitted 2024-02-15; First posted 2024-03-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cytomegalovirus Infection
Keywords: Cytomegalovirus infection; Cytomegalovirus disease
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir; Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letermovir+Valganciclovir (Experimental): Daily administration of Letermovir plus Valganciclovir
  Interventions: Drug: Letermovir; Drug: Valganciclovir
- Letermovir Placebo+Valganciclovir (Active Comparator): Daily administration of Letermovir placebo plus Valganciclovir
  Interventions: Drug: Valganciclovir; Drug: Letermovir placebo

INTERVENTIONS:
Drug: Letermovir — 480mg (2X240mg- tablets) of Letermovir given orally once a day until the "treatment success" or the "treatment failure", up to 12 weeks. In case of co-administration with cyclosporine A, the dosage of Letermovir will be reduced.
  Arms: Letermovir+Valganciclovir
Drug: Valganciclovir — Valganciclovir 900 mg (2X450 mg-tablets) twice a day until the "treatment success" or the "treatment failure", up to 12 weeks. In case of impaired renal function, the dosage of valganciclovir will be reduced.
Drug: Letermovir placebo — 480mg (2X240mg- tablets) of Letermovir placebo given orally once a day until the "treatment success" or the "treatment failure", up to 12 weeks
  Arms: Letermovir Placebo+Valganciclovir

SUMMARY:
The purpose of this study is to evaluate the efficacy and the tolerance of letermovir as part of dual antiviral therapy (in association with valganciclovir) in renal transplant recipients with CMV DNAemia, requiring valganciclovir treatment per investigator's judgment.

DETAILED DESCRIPTION:
Ganciclovir and valganciclovir are the drugs of choice to treat CMV infections and diseases in immunocompromised patients. However, (val)ganciclovir does not seem to be a panacea and its modest efficacy and dose-limiting toxicities limit effectiveness. More, (val)ganciclovir use may drive development of drug-resistant infections, particularly in immunocompromised patients.

An in vitro study suggested additive effects for the combination of letermovir with all approved drugs for treatment or prevention of CMV infections. Investigator's hypothesis is that letermovir plus valganciclovir dual therapy will inhibit CMV replication faster than valganciclovir monotherapy. More, the use of antiviral dual therapy aims to decrease the risk of drug resistance mutations' selection, as previously demonstrated in several other viral infections.

In this study, renal transplant recipients with CMV DNAemia requiring valganciclovir will be randomized to receive either letermovir plus valganciclovir or letermovir placebo plus valganciclovir, until reaching the "treatment success" or the "treatment failure" criteria, up to 12 weeks.

Treatment success will be defined as, from Week-3:

* eradication of CMV DNAemia, defined as CMV DNAemia in whole blood below lower limit of quantification (LLOQ) < 200 IU/mL on 1 blood sample.
* AND resolution of clinical symptoms of CMV disease (if appropriate)

Treatment failure will be defined as fulfilling at least one criterion among:

* failure to achieve a decrease of CMV DNAemia ≥ 1 log10 IU/mL at Week-3 compared to the baseline CMV DNAemia
* persistence of CMV DNAemia ≥ LLOQ (200 IU/ml) at Week-12
* absence of improved CMV disease at Week-3.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Weight ≥ 30 kg
3. Kidney transplant recipient
4. Have a documented CMV infection or disease, with (i) a screening value of CMV DNA ≥ 3000 IU/mL in whole blood or plasma in 2 consecutive assessments separated by ≥ 1 day, as determined by local laboratory quantitative polymerase chain reaction (qPCR). Both samples should be taken within 14 days prior to randomization with the second sample obtained within 5 days prior to randomization OR (ii) a screening value of CMV DNA ≥ 30000 IU/mL in whole blood or plasma, as determined by local laboratory quantitative polymerase chain reaction (qPCR), in 1 sample obtained within 5 days prior to randomization
5. Eligible for treatment with oral valganciclovir, per investigator's judgment
6. For patients of childbearing age (following menarche): negative bHCG and effective method of contraception (sexual abstinence, hormonal contraception containing ethinylestradiol and levonorgestrel, intrauterine device or hormone-releasing system, cap, diaphragm or sponge with spermicide, condom) until 30 days after the end of relevant systemic exposure (week 13).

   For male an effective method of contraception (sexual abstinence, condom) until 90 days after the end of relevant systemic exposure (week 13).
7. Have life expectancy of ≥ 8 weeks
8. French speaking
9. Affiliated to social security regime or an equivalent system
10. Informed consent and signed

Exclusion Criteria:

1. Have a current CMV infection that is considered refractory or resistant due to inadequate adherence to antiviral treatment, to the best knowledge of the investigator.
2. Have a CMV infection that is known to be genotypically resistant to valganciclovir and/or letermovir on documented evidence.
3. Be on treatment with anti-CMV agents (ganciclovir, valganciclovir, foscarnet, cidofovir, letermovir or maribavir) for the current CMV infection for longer than 72 hours. However, patients experiencing CMV infection while receiving ganciclovir or valganciclovir prophylaxis (i.e. at prophylactic dosages) or letermovir prophylaxis can be included.
4. Have an eGFR < 15 mL/min/1.73m² (using the CKD-EPI Creatinine Equation (2009)).
5. Have serum aspartate aminotransferase (AST) ≥ 5 times higher than the upper limit of normal (ULN), or serum alanine aminotransferase (ALT) ≥ 5 times the ULN, or total bilirubin ≥ 3 times the ULN (except for documented Gilbert's syndrome). Note: Subjects with biopsy confirmed CMV hepatitis will not be excluded from study participation despite AST or ALT ≥ 5 times ULN
6. Have a severe chronic liver disease (Child-Pugh Class C)
7. Have a known human immunodeficiency virus (HIV) infection with plasma HIV RNA ≥ 50 copies/mL within the 3 months before inclusion.
8. Require mechanical ventilation or vasopressors for hemodynamic support.
9. Be pregnant or breastfeeding.
10. Have received anti-CMV vaccine at any time.
11. Be receiving leflunomide or artesunate when study treatment is initiated.
12. Be receiving strong inhibitors or inducers of hepatic CYP enzymes including rifampicin, phenytoin, clarithromycin, ritonavir, or cobicistat or St. John's wort (Hypericum perforatum) when study treatment is initiated.
13. Be receiving efavirenz, etravirine, nevirapine, lopinavir, pimozine, ergot alkaloids, dabigatran, atorvastatine (at a daily dose > 20mg, and / or if co-administered with cyclosporin A), pravastatin ( if co-administered with cyclosporin A), simvastatine, rosuvastatine, pitavastatine or imipenem-cilastatine when study treatment is initiated.
14. Have known hereditary intolerance to galactose, with lactose Lapp deficiency, glucose or galactose malabsorption syndrome.
15. Have known hypersensitivity to letermovir or to an excipient for a study treatment.
16. Have any clinically significant medical or surgical condition that in the investigator's opinion could interfere with the interpretation of study results, contraindicate the administration of the assigned study treatment, or compromise the safety or well-being of the subject.
17. Participation to another clinical trial on medicinal products for human use
18. Have an absolute neutrophil count less than 500 cells/µl, or platelet count less than 25,000/µl, or haemoglobin less than 8 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Virological response to treatment on week-3 | 3 weeks
  defined as a ≥ 2 log10 decrease of CMV DNAemia in whole blood from baseline, or an undetectable CMV DNAemia (< 200 IU/mL) in whole blood

SECONDARY OUTCOMES:
Eradication of CMV DNAemia (< 200 IU/ml) before Week-12 | 12 weeks
  quantitative CMV PCR performed in whole blood every week until interruption of antiviral treatment, or at the latest until Week-12
Number of days between baseline and first measure of CMV DNAemia < 200 IU/mL | 12 weeks
  Quantitative CMV PCR performed in whole blood every week until interruption of antiviral treatment, or at the latest until Week-12
Absence of CMV-related disease or syndrome at baseline and each visit | 12 weeks
Adverse event (AE) occurence | 12 weeks
  Clinical examination and clinical laboratory assessments performed every week until interruption of antiviral treatment (or at the latest until Week-12)
Sequencing of whole UL97, UL54, UL56, UL89 and UL51 genes | 12 weeks
  in blood samples at baseline, at Week-3 or Week-12 (in patients achieving criteria defining "treatment failure"), and at any visit in patients presented with rebound of CMV DNAemia
Ganciclovir plasma concentration | 2 weeks
  at Week-1 and Week-2, in case of premature termination of treatment for any reason or premature exit from the study.
Letermovir plasma concentration | 2 weeks
  t Week-1 and Week-2, in case of premature termination of treatment for any reason or premature exit from the study.
Measure of the CMV specific T-cell immunity | 12 weeks
  at baseline, Week-3, Week-6, Week-9 and Week-12.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne LERUEZ-VILLE, MD, PhD, Study Chair — Virology laboratory- reference national Lab for CMV infection -Hôpital Necker Enfants malades, Paris; Pierre FRANGE, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux Paris
Locations (5):
- France (5):
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital de la Pitié Salpêtrière, Service de Néphrologie, Paris, Île-de-France Region
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region
  - Hôpital Necker Enfants Malades - SMIT, Paris, Île-de-France Region
  - Centre 011-Hôpital Bichat, Service de Néphrologie, Paris, Île-de-France Region